CLINICAL TRIAL: NCT03829982
Title: The Effects of Light on Glucose Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Collaborators: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NL63655.068.17
Record Dates: First submitted 2019-01-10; First posted 2019-02-04 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Diabetes Mellitus, Type 2; Glucose Intolerance; Prediabetic State
Keywords: Circadian Rhythm
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance; Prediabetic State

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bright light during the day (Experimental): Participants will be exposed to bright light (1250 lux) between 8:00 and 18:00 and to dim light (5 lux) between 18:00 and 23:00.
  Interventions: Behavioral: Exposure to bright light during the day
- dim light during the day (Experimental): Participants will be exposed to dim light (10 lux) between 8:00 and 18:00 and to dim light (1250 lux) between 18:00 and 23:00.
  Interventions: Behavioral: Exposure to dim light during the day

INTERVENTIONS:
Behavioral: Exposure to bright light during the day — Participants will be exposed to bright light (1250 lux) between 8:00 and 18:00 and to dim light (5 lux) between 18:00 and 23:00.
  Arms: bright light during the day
Behavioral: Exposure to dim light during the day — Participants will be exposed to dim light (10 lux) between 8:00 and 18:00 and to dim light (1250 lux) between 18:00 and 23:00.
  Arms: dim light during the day

SUMMARY:
This study evaluates the effect of bright light on postprandial blood glucose metabolism in obese subjects with impaired fasting glucose and/or impaired glucose tolerance.

DETAILED DESCRIPTION:
Light has a major influence on the biological clock and several studies suggest that bright light during the day and dim light in the evening are beneficial for the circadian timing system. Nowadays, large parts of the population spend 90% of their time indoors and are thereby exposed to artificial lighting instead of daylight. The artificial light levels are relatively low during the day and continue relatively late in the evening. The lack of a clear natural light-dark cycle could results in delayed timing of the biological clock relative to the behaviour. Optimizing the lighting conditions under controlled laboratory settings might lead to better alignment of the biological clock, which in turn could improve metabolic parameters such as glucose control.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* BMI 25-35 kg/m2
* Stable weight (+/- 3 kg in the last 3 months)
* One of the four criteria for prediabetes:

  * Impaired fasting glucose (6.1 mM to 6.9 mM)
  * Blood glucose values 7.8 - 11.1 mM 2h after glucose drink consumption during the oral glucose tolerance test (OGTT) in screening
  * Insulin Resistance: glucose clearance rate ≤ 360 ml/kg/min, as determined using the oral glucose insulin sensitivity (OGIS120) index
  * HbA1c of 5.7 - 6.4%.

Exclusion Criteria:

* Fasting plasma glucose ≥7.0 mM
* Blood donation one month prior to study and three months after finishing study.
* Participants with extreme chronotypes (going to bed extremely late/early).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
Postprandial glucose (mg/dL) | Study Day 1-3
  Assessed with a continuous glucose monitor (CGM)

SECONDARY OUTCOMES:
Glucose levels (mmol/L) in the postprandial state | Study Day 2-3
  venous blood draw every 30 min for 4 hours after breakfast and after dinner
Free fatty acid levels (µmol/L) in the postprandial state | Study Day 2-3
  venous blood draw every 30 min for 4 hours after breakfast and after dinner
Triglycerides levels (mmol/L) in the postprandial state | Study Day 2-3
  venous blood draw every 30 min for 4 hours after breakfast and after dinner
Insulin levels (µU/mL) in the postprandial state | Study Day 2-3
  venous blood draw every 30 min for 4 hours after breakfast and after dinner
Continuous interstitial glucose (mg/dL) | Study Day 1-3
  Assessed with continuous glucose monitor (CGM)
Energy expenditure | Study Day 1-3
  continuous measurement with whole room indirect calorimetry
Core body temperature (CBT) and skin temperature | Study Day 1-3
  Measured with a telemetric pill (CBT) and 14 temperature sensors (iButtons) in degrees celsius

CONTACTS AND LOCATIONS:
Overall Officials: Wouter van Marken Lichtenbelt, Prof. Dr., Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Harmsen JF, Wefers J, Doligkeit D, Schlangen L, Dautzenberg B, Rense P, van Moorsel D, Hoeks J, Moonen-Kornips E, Gordijn MCM, van Marken Lichtenbelt WD, Schrauwen P. The influence of bright and dim light on substrate metabolism, energy expenditure and thermoregulation in insulin-resistant individuals depends on time of day. Diabetologia. 2022 Apr;65(4):721-732. doi: 10.1007/s00125-021-05643-9. Epub 2022 Feb 2. PMID 35106618